CLINICAL TRIAL: NCT06258655
Title: The Change Mechanisms of the Close Collaboration With Parents Intervention and the Adaptability of the Intervention in the Estonian Context
Brief Title: The Effect of the Close Collaboration With Parents Intervention - Estonian Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: University of Tartu (Other)
Responsible Party: Principal Investigator, Sari Ahlqvist-Bjorkroth, Associate Professor, University of Turku
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: SA332962
Record Dates: First submitted 2023-02-03; First posted 2024-02-14 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Depression, Postpartum; Anxiety
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A quasi-experimental before and after intervention design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (No Intervention): The sample collected before the intervention
- Post-intervention (Experimental): The sample collected after the intervention
  Interventions: Other: Close Collaboration with Parents

INTERVENTIONS:
Other: Close Collaboration with Parents — The Close Collaboration with Parents intervention is an educational program for the neonatal staff to improve their skills to collaborate with parents and provide support to parenting during an infant's hospitalization. First, experienced nurses and doctors from the units will undergo a 14-day to become "unit mentors". Then these unit mentors will train other members of staff. The training of the units is based on bedside practices, a reflection of the practices, and the application of the knowledge in everyday work. Theoretical learning, preceding clinical bedside mentoring, will occur through an e-learning module. Staff members will spend about 4 working days in training alongside their routine work. The unit mentors will function as facilitators for the staff, and they have dedicated time for this. The content of the bedside practices is guided by a manual. The training team will provide frequent remote and contact support for the implementation.
  Arms: Post-intervention

SUMMARY:
The overall aim of the study is to implement an evidence-based intervention called 'Close Collaboration with Parents' in Estonian neonatal units. The goal of the intervention is to educate the whole multi-professional NICU staff and promote a positive change in the family-centered care culture of the units. Thus, the first aim of the study is to implement the intervention in an Estonian NICU context, in three hospitals, and study the fidelity of the intervention. More precisely, the study questions are whether adaptations are needed for the successful implementation of the intervention in the Estonian context and how feasible are the used implementation strategies. Secondly, the aim is to study the effectiveness of the Close Collaboration with Parents intervention in this context by using a quasi-experimental, pre-test - post-test, study design. The questions are whether the implementation of the intervention in the Estonian setting will result in positive effects such as 1) an improved development environment for the infants during hospital stay (less noise, more parental speech, and more parent-infant physical closeness), 2) intensified parental bonding to the infant, and 3) increased parental confidence and emotional well-being at the time of discharge from hospital.

DETAILED DESCRIPTION:
Materials and Methods: Design A quasi-experimental, before and after intervention, design is used to test the effect of the intervention, where the impact mechanisms are treated as mediators of the change.

Sample: The subjects are employees of five neonatal units of three Estonian hospitals participating in the Close Collaboration with Parents intervention (hereinafter: staff) and newborns cared for in the units and their parents (hereinafter: families). Three of the units are at Tallinn: West-Tallinn Maternity Hospital (NICU and neonatal unit), the Department of Anesthesiology and Intensive Care (PICU/level IIIB), and the Department of Neonatal and Infant Medicine (NICU/level II) at the Children's Hospital. Another two units are located in Tartu University Hospital: the Department of Neonatal and Pediatric Intensive Care (PNICU, level IIIC) and a step-down unit (level II).

Families are recruited during a four-month period before and after the intervention, with the aim to recruit at least 50 families per participating hospital in both periods. Some newborns may be treated in a different hospital or in different units of the same hospital. In the case of a transfer, the family is asked to fill in only the Family Center questionnaire if the newborn has been in that unit for more than 72 hours.

A log will be kept of all infants discharged home from the unit i.e. to evaluate drop-out rate and biases. The log includes the patient's gestational age, birth weight, diagnosis, type of feeding at discharge, and length of hospital stay. If there is missing information in the log, it is completed with the information from the medical records. A log is also kept to follow the units' restrictions related to Covid-19 and concerning family visitation and participation policies.

Outcomes:

The fidelity is analyzed by tracking the participants' behavior in the e-learning module with analytic software, such as Google Analytics, Hotjar, and Vimeo. The participants are informed about this and they are asked for their written consent and agreement when entering the module for the first time. Furthermore, a log is kept about the practices the mentors are carrying out with their colleagues in the units.

Staff outcomes Background questionnaire A questionnaire is used to collect background information on staff members Collaboration competence questionnaire A questionnaire is used to assess the collaboration competence of the staff at the beginning of the intervention, in the middle of the implementation, and at the end. The questionnaire is specifically created to assess competencies that are relevant to the Close Collaboration with Parents training program. The questionnaire includes 21 questions that are evaluated with a scale from 1 to 10 (1=not competent at all, 10=extremely competent). If the question does notably the daily work role of the professional option, "Doesn't belong to my role" can be used.

The reflective thinking The level of reflective thinking of the staff is measured using the Reflective Thinking Measure. The 16-question measure determines whether an individual engages in reflective thinking and to what extent s/he does that. The questions are answered with options varying from strongly agree, which is scored as 5, to strongly disagree, which is scored as 1. The 16 questions form four factors: 1) Habitual Actions, 2) Understanding, 3) Reflection, and 4) Critical reflection. The structural validity of the scale has been tested on healthcare professionals and it has been shown to be good.

The level of reflective thinking is also assessed with questions related to a fictitious case. The case represents a so-called 'critical incident' that the staff is asked to describe from three perspectives: (a) how they would normally act in a similar situation in their unit; (b) a general meaning and reflect how the general meaning resonates with their own experience; and (c) potential new ways of acting in the situation that would provide better support for the family The FCC care provision The perception of multi-professional staff members on parent support they have given that day is measured with DigiFCC web questions. The question will reflect the staff's point of view on the support provided for parents in the following dimensions: 1) active listening, 2) parent participation in infant care, 3) individualized parent education, 4) parent participation in decision-making, 5) the parent trust staff in infant care, 6) the staff feel the parents trust them in infant care, 7) participation in medical round/medical care decision making, 8) information sharing, and 9) emotional support. Staff members answer the questions through a website that is always open on the research computer in the unit. Every staff member (regardless of qualifications) working in the participating units is asked to answer a daily question through a website after each work shifts for a 3-month period. There are 9 questions that are randomized in 3-question blocks. Answers are numbers from 1 to 5 or 0 if the staff member hasn't been working with the parents on that shift or didn't participate in the medical round.

Regarding the same 4-month period, the researcher/administrator collects the number of nursing staff working shifts in the unit to calculate the response rate. The research will create a questionnaire for each unit through the Master account website. The responsible researcher will have access to the research account to collect the answers.

Family outcomes Infant-parent background questionnaire A questionnaire is used to collect background information on infants/parents Parents' depressive symptoms The depressive symptoms of parents are measured with Edinburgh Postnatal Depression Scale (EPDS). The 10-question EPDS is a valid method to measure depressive symptoms both in mothers and fathers. The 10-question scale includes symptoms such as insomnia, mood, tearfulness, and thoughts of self-harm. The scale asks how the parent has felt during the previous week. The parents rate each question on a scale from 0 to 3. The EPDS is easy to administer and has high sensitivity as a screening tool.

Parent's anxiety symptoms The anxiety symptoms of the parents are assessed with State and Trait Anxiety Inventory (STAI). State anxiety is an emotional reaction that varies from one situation to another, whereas trait anxiety is a personality characteristic. The STAI measurement provides separate scores for both types of anxiety. There are 20 questions about state anxiety that are rated with a 4-point scale (1=not at all, 4=very much) and 20 questions about trait anxiety that are also rated with a 4-point scale (1=almost never, 4=almost always). The recommended cut-off for postnatal anxiety measured with STAI-S is 34/80.

The research assistant will calculate the parent's scores of EPDS and STAI-S when the questionnaires are returned. She informs the responsible researcher of the unit if the total score of the EPDS is >12 or if the parent has suicidal thoughts and if the total score of STAI-S is >33.

Parenting self-efficacy scale Parenting self-efficacy is measured Perceived Maternal Parenting Self-Efficacy (PMP S-E) instrument. The PMP S-E instrument consists of 20 items (scoring ranges 20-80) with four subscales: 1) care-taking procedures, 2) evoking behaviors, 3) reading behaviors or signaling, and 4) situational beliefs. The items are rated with a four-point Likert scale ranging from 'strongly disagree' (score 1) to 'strongly agree' (score 4). The PMP S-E tool is a psychometrically robust, reliable, and valid measure of parenting self-efficacy in mothers of relatively healthy hospitalized preterm neonates.

Parent's readiness for discharge The readiness for discharge is measured with the Readiness for Hospital Discharge Scale (RHDS). The questionnaire includes 23 items. Four attributes of readiness for discharge are measured within the subscales: Personal Status (7 items), Knowledge (7 items), Coping Ability (4 items), and Expected Support (5 items). Answers are on a 10-point scale from 0 to 10 (not at all - totally). The RHDS has been shown to be a reliable and valid measure of patients' perception of readiness for discharge.

Parent's perceived FCC The parent participation and the support parents feel they receive from the staff is measured using a questionnaire modified from DigFCC SMS questions. The questionnaire includes 9 questions covering the following aspects of staff support 1) active listening, 2) parent participation in infant care, 3) individualized parent education, 4) parent participation in decision-making, 5) the parent trust staff in infant care, 6) the parent feel the staff trust them in infant care, 7) participation in medical round/medical care decision making, 8) received information, and 9) emotional support. They are asked to answer the question with the Likert scale from 1 to 7 (1=not at all-7=very much; 0= if they did not visit the unit).

Data management The investigators will utilize REDcap (Research Electronic Data Capture) for data transfers from Estonia to Finland and for data storage. REDcap is an electronic tool for data collection that is provided from the server facilities owned and operated by the University of Turku IT Services, which also means all data collected to the system is stored and kept at the University of Turku. When the data is stored in the online file storage of Turku University it is automatically copied to three independent servers that also function as data backup systems.

Data security description:

* Centralized administration by separate administration accounts and compartmentalized user privileges
* Use of current and reliable hardware, and software which is updated continuously
* Centralized identity management (IDM)
* Locally administered industry-standard network infrastructure and services
* Common server platforms with minimal tailoring
* Continuous monitoring of network traffic patterns and service statistics
* Widely deployed security software and other monitoring tools The principal investigator (PI) controls access to the data. The co-researchers can approach the PI to request access to the data. The PI will apply to the University of Turku IT Services to provide the access to the online storage. If a co-researcher is not working at the University of Turku, the PI can ask the IT services to give that person a visitor status and, thereby, access to the online file storage. All new users are identified using government-issued identification documents or by citizens' identification and payment service. The IP will keep a record of those who have active access to the data.

All the data will be handled anonymously. The participants will get an ID code that is used when data is stored and analyzed. The recruitment log of the parents and staff members are used to undo the ID codes and, therefore, they are kept separately from the data files. The analytic software (Google Analytics, Hotjar, and Vimeo) also track anonymously participants' behavior on the e-learning module's website. The personal details (password, email, etc) are not recorded and the IP addresses are anonymized by cutting out the last few digits, so only the rough geographical area of access to the e-learning module is identified. The logs and all the data will be destroyed five years after the last publication of the data.

Ethical considerations Ethical approval for the study protocol was given by the Research Ethics Committee of the University of Tartu on the 10th of February 2021 (no: 3331T-21). Written informed consent will be obtained from each staff member and parent before study participation. The analytic software (Google Analytics, Hotjar, and Vimeo) will be activated only after consent has been obtained from a participant. The application for ethics includes an opportunity to complete the information received from the parents (infant and family characteristics questionnaire) using patient medical records.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the families are:

1. families whose newborns have been hospitalized during the first 28 days of infant life
2. expected length of stay of the newborn is at least three days
3. discharge is planned to happen within a week
4. at least one parent has agreed to participate in the study

The exclusion criterion for the families:

1) Not able to communicate in Estonian, Russian, or English.

The inclusion criterion for the staff members:

1) The staff working in the units during the entire study period are eligible for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Depression | Up to 2 months
  The postnatal depressive symptoms of the mothers whose newborn has been cared for in the unit after the intervention are compared with the postnatal depressive symptoms of the mothers whose newborn has been cared for in the unit before the intervention. The symptoms are measured with Edinburgh Postnatal Depression Scale. The 10-question scale includes symptoms such as insomnia, mood, tearfulness, and thoughts of self-harm. The scale asks how a person has felt during the previous week. The minimum score is 0 and the maximum is 30. A high score indicates more depressive symptoms.

SECONDARY OUTCOMES:
Anxiety | Up to 2 months
  The measurement provides separate scores for both state and trait anxiety. There are 20 questions about state anxiety with a minimum score of 20 and a maximum of 80 and 20 questions about trait anxiety with the same minimum and maximum scores. A high score indicates more anxiety symptoms.

OTHER OUTCOMES:
Parenting self-efficacy | Up to 2 months
  Parenting self-efficacy is measured using the Perceived Maternal Parenting Self-Efficacy questionnaire. The questionnaire consists of 20 items. The total score on the scale ranges from 20 to 80. A high score indicates more parenting self-efficacy.
Readiness for discharge | Up to 2 months
  The readiness for discharge is measured with the Readiness for Hospital Discharge Scale. The questionnaire includes 23 items. The total score on the scale ranges from 0 to 230. A high score indicates more readiness for discharge.
Family-centered care | Up to 2 months
  The parent participation and the support parents feel they receive from the staff are measured using a questionnaire modified from Digital Family-Centered Care questions that were made for the Short Message Service. The questionnaire includes 9 items. The total score on the scale ranges from 7 to 49. A high score indicates more that the received care is experienced as more family-centered.
Reflective thinking | Through study completion, an average of 2 years and 2 months
  The level of reflective thinking of the staff is measured using the Reflective Thinking Measure. The 16-question measure determines whether an individual engages in reflective thinking and to what extent s/he does that. Scores range from 16 to 80, with 80 indicating the highest possible level of reflection.

CONTACTS AND LOCATIONS:
Overall Officials: Sari Ahlqvist-Björkroth, Assoc.Prof., Principal Investigator — University of Turku; Heili Varendi, Prof., Study Director — University of Tartu and Tartu University Hospital; Liis Toome, MD, Study Chair — Tallinn Children's Hospital; Pille Saik, MD, Study Chair — West Tallinn Central Hospital; Liisa Lehtonen, Prof., Study Director — University of Turku
Locations (1):
- Sari Ahlqvist-Björkroth, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
Because data includes sensitive information about the patients we are not planning to share individual participant data (IPD). However, the study protocol, statistical analysis plan, and used informed consent forms can be shared. The results of the study are shared in study reports in research journals.

REFERENCES:
- [Derived] Itoshima R, Varendi H, Toome L, Saik P, Axelin A, Lehtonen L, Moazami-Goodarzi A, Ahlqvist-Bjorkroth S. Outcomes Following Close Collaboration With Parents Intervention in Neonatal Intensive Care Units: A Nonrandomized Clinical Trial. JAMA Netw Open. 2025 Jan 2;8(1):e2454099. doi: 10.1001/jamanetworkopen.2024.54099. PMID 39786771
- See also: e-learning tool used in the intervention — https://closecollaboration.utu.fi/